CLINICAL TRIAL: NCT07112131
Title: The Effect of Non-Diet Nutrition Education on Eating Behavior, Body Image, and Well-Being in Adult Women: A Randomized Controlled Trial
Brief Title: Non-Diet Nutrition Education and Its Effects on Eating Behavior, Body Image, and Well-Being in Adult Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba TÜRKCAN (Other)
Responsible Party: Sponsor-Investigator, Tuğba TÜRKCAN, Principal Investigator, Istanbul Gelisim University
Organization: Istanbul Gelisim University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KA23/243
Record Dates: First submitted 2025-07-16; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Eating Behaviors; Body Image; Well-Being, Psychological; Young Adult Females
Keywords: Non-diet approach; Intuitive eating; Body acceptance; Body image; Eating behavior; Psychological well-being; Young adult women; Nutrition education; Randomized controlled trial
MeSH Terms: conditions — Feeding Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group receiving an 8-week online non-diet nutrition education program or a control group receiving no intervention.
Who Masked: Participant
Masking Description: Participants are blind to the group assignment and the primary aim of the study. The study is designed as a single-blind randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive an 8-week online non-diet nutrition education program based on intuitive eating and body acceptance principles.
  Interventions: Behavioral: Non-Diet Nutrition Education Program
- Control Group (No Intervention): Participants in this group will receive no intervention during the 8-week study period but will complete the same pre- and post-assessments as the intervention group.

INTERVENTIONS:
Behavioral: Non-Diet Nutrition Education Program — The intervention is an 8-week online nutrition education program based on non-diet approaches, including intuitive eating, rejecting diet mentality, honoring hunger, body acceptance, and well-being. Each weekly session is 60 minutes long and involves interactive discussions and home practices.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a non-diet nutrition education program can improve eating behaviors, body image, and well-being in normal-BMI women aged 19-35 years. The main questions it aims to answer are:

* Does participation in an 8-week non-diet nutrition education program improve eating behavior, body image, and well-being over time in the intervention group compared to the control group?
* Is there a significant difference between the intervention and control groups in eating behavior, body image, and well-being after the intervention?

Researchers will compare an intervention group receiving an 8-week non-diet nutrition education with a control group receiving no intervention, to see if the program leads to improvements in psychological and behavioral outcomes without focusing on weight loss.

Participants will:

* Complete pre- and post-intervention assessments, including validated questionnaires on eating behavior (DEBQ, FCQ, IES-2), body image (BAS, Stunkard Figure Rating Scale), and psychological well-being (WHO-5, Rosenberg Self-Esteem Scale), as well as a 3-day food diary.
* Be randomly assigned to either the intervention group (8-week online non-diet nutrition education sessions) or the control group (no intervention).
* Engage in 8 weekly, 60-minute sessions focused on intuitive eating, body acceptance, and health-promoting nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Aged between 19-35 years,
* Body Mass Index (BMI) between 18.5-24.9,

Exclusion Criteria:

* Pregnant or breastfeeding,
* Diagnosed eating disorder or other psychiatric condition,
* Currently enrolled in a weight loss program,
* Following a restrictive diet due to medical conditions.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Eating Behavior | Baseline and 8 weeks after intervention
  Assessed using the Dutch Eating Behavior Questionnaire (DEBQ): 33 items with three subscales (Restrained Eating, Emotional Eating, External Eating), rated on a 5-point Likert scale (1 = never, 5 = very often). Higher subscale scores indicate greater tendency toward that eating behavior.
Food Choice Motivation | Baseline and 8 weeks after intervention
  Assessed using the Food Choice Questionnaire (FCQ): 36 items, 9 subscales (Health, Mood, Convenience, Sensory Appeal, Natural Content, Price, Weight Control, Familiarity, Ethical Concern), rated on a 4-point Likert scale (1 = not at all important, 4 = very important). Higher scores indicate greater importance assigned to that factor in food choice.
Intuitive Eating | Baseline and 8 weeks after intervention
  Assessed using the Intuitive Eating Scale-2 (IES-2): 23 items, 4 subscales (Unconditional Permission to Eat, Eating for Physical Rather Than Emotional Reasons, Reliance on Hunger and Satiety Cues, Body-Food Choice Congruence), rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores reflect more intuitive eating.
Body Appreciation | Baseline and 8 weeks after intervention
  Assessed using the Body Appreciation Scale (BAS): 9 items, no subscales, rated on a 5-point Likert scale (1 = never, 5 = always). Higher scores indicate greater body appreciation.
Body Dissatisfaction | Baseline and 8 weeks after intervention
  Assessed using the Stunkard Figure Rating Scale: visual selection of perceived vs. ideal body silhouette (1-9 scale). Body dissatisfaction is calculated as the difference between the actual and ideal figure selections.
Well-Being | Baseline and 8 weeks after intervention
  Assessed using the WHO-5 Well-Being Index: 5 items, no subscales, scored 0-5 (0 = at no time, 5 = all the time); raw scores are converted to a 0-100 scale. Higher scores indicate better well-being.
Self-Esteem | Baseline and 8 weeks after intervention
  Assessed using the Rosenberg Self-Esteem Scale (RSES): 10 items, no subscales, rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Higher scores reflect greater self-esteem.

SECONDARY OUTCOMES:
Dietary Intake | Baseline and 8 weeks after intervention
  Description:
  Assessed via 3-day food record (2 weekdays and 1 weekend day). Food items are recorded by participants using visual portion guides. Analysis performed using eBebis (Turkish Nutrition Database software).
  Unit of Measure:
  * Energy intake (kilocalories/day)
  * Macronutrient intake (grams/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including questionnaire responses (e.g., DEBQ, FCQ, IES-2, WHO-5), will be available to qualified researchers for academic and non-commercial use upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting information will be available starting 6 months after publication of the main study results and will remain available for up to 3 years upon request.
Access Criteria: IPD and supporting documents will be made available to qualified researchers with a valid academic affiliation. Access will be granted upon submission of a research proposal and a data use agreement. Requests should be directed to the principal investigator via institutional email.